CLINICAL TRIAL: NCT07023406
Title: Effectiveness of and Implementation Strategies for 'Disfrutando': A Culturally Tailored, Bundled Intervention to Address Type 2 Diabetes Mellitus in High-burden Populations
Brief Title: Effectiveness of and Implementation Strategies for 'Disfrutando'.
Acronym: Disfrutando 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Maithe Enriquez, Professor in Nursing, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0082846
Record Dates: First submitted 2025-05-29; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Participatory Research; T2DM; High-Burden Populations
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, waitlisted, design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Behavioral Intervention
  Interventions: Behavioral: Disfrutando
- Waitlist Group (Experimental): This arm will receive the intervention after the waitlist period
  Interventions: Behavioral: Disfrutando

INTERVENTIONS:
Behavioral: Disfrutando — Disfrutando is a six-week, weekly intervention with a booster intervention at week 12. Intervention content includes glucose control with individual goals, glucose monitoring and glucometer practice, healthy eating demonstrations, benefits of physical activity, prevention and management of T2DM. The intervention has a strong focus on mitigating barriers and challenges to diabetes self-care management.

SUMMARY:
Despite much research that has focused on enhancing type 2 diabetes mellitus (T2DM) health outcomes for high burden populations, more remains to be done. There is a need to develop practical approaches that not only equip people with knowledge about T2DM self-management, but also help them mitigate the adverse social determinants of health (SDOH) that are fueling the burgeoning numbers of people in the United States with T2DM and that are preventing them from practicing healthful behaviors. This study will examine an intervention named 'Disfrutando' that strives to help people prevent and manage T2DM.

DETAILED DESCRIPTION:
The investigators have engaged a community-health-academic partnership that is working to move a program of research forward that addresses the 'epidemic' of T2DM in high burden populations in Missouri. The partnership developed the Disfrutando intervention in a non-controlled feasibility study with encouraging results: Hemoglobin A1C (i.e., average blood sugar levels) was lowered for 66% of 31 participants. Disfrutando is an interactive, culturally tailored, bundled intervention that aims to enhance self-efficacy and equip people with knowledge and skills about healthful behaviors (i.e., healthy eating, physical activity) and engage them in primary/diabetes/eye care to enhance diabetes health outcomes. What makes Disfrutando stand out is its facilitation by community health workers who focus on "meeting people where they are" and connecting them to no- or low-cost resources that increase access to/engagement in healthy eating, physical activity, and primary/diabetes/eye care. The investigators now propose a 1-year pilot study that will examine the effectiveness of and implementation strategies for Disfrutando using a two-group randomized, wait-list controlled design. Hypotheses are: (1) implementation quality and acceptability of the Disfrutando intervention will be high and (2) the intervention will lower HbA1C, change body weight, enhance self-efficacy, and mitigate adverse SDOH. Research Questions are: RQ1: What is the implementation quality of the intervention? (i.e., adherence to intervention content, characteristics of intervention delivery), RQ2: Are people engaged and satisfied with the intervention?, RQ3: What is the impact of Disfrutando on HbA1C and change in body weight?, and RQ4: What is the relationship between HbA1C, change in body weight and selected mediators (diabetes self-efficacy, quality of intervention delivery, mitigation of SDOH (i.e., access and linkage to resources for engagement in healthy eating, physical activity, and attendance at health care appointments) and moderators (personal and health characteristics)? This pilot project will provide critical effectiveness and implementation data to inform an application for a multi-site community trial. Early identification and management of pre-diabetes and T2DM is critical for the prevention of diabetes-related serious health problems and premature death.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin A1C of 5.7 or higher

Exclusion Criteria:

* Hemoglobin A1C of 5.6 or lower

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glucose (Blood Sugar) Control | Hemoglobin A1C will be measured at baseline (pre-intervention), 12 weeks, and 6 months.
  Name of measurement: Hemoglobin A1c (HbA1C) How measured/assessed: HbA1C is a biomedical test that provides average glucose (blood sugar) level over the past 8 to 12 weeks and is used to help manage diabetes. Glucose (blood sugar) control will be evaluated using the A1CNow Self Check device. This FDA-cleared device is sold over the counter and is a portable, self-check test that is self-administered using a small fingerstick blood sample. Results are obtained in 5 minutes.

SECONDARY OUTCOMES:
Change in Body Weight | Body weight will be measured weekly for 6 weeks, at 12 weeks, and at 6 months. The same scale will be used at all time points.
  Name of Measurement: Change in Body Weight. How measured/assessed: weight will be measured using a medical-grade scale. Weight is a modifiable contributor to type 2 diabetes mellitus (T2DM), and addressing overweight can enhance T2DM health outcomes.
Self-efficacy for diabetes self-care management | Self-efficacy will be measured at pre-intervention, 12 weeks, and 6 months
  Name of measurement: Diabetes Self-Efficacy Scale. How measured/assessed: Self-efficacy is hypothesized as a mediator of engagement in healthful diabetes-related behaviors. Self-efficacy (i.e., confidence that an individual has for managing their diabetes) will be measured with the Diabetes Self-Efficacy Scale, a questionnaire with 8 questions that was developed by the Stanford Patient Education Center. The questionnaire uses a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident) in the ability to perform activities to manage diabetes, such as diet, exercise, and following up with healthcare providers.